CLINICAL TRIAL: NCT03429920
Title: The Effect of Fermented Soy Based Dietary Food Product on Cardiometabolic Risk Factors in Individuals at High Risk of Cardiovascular Disease
Brief Title: Effect of Fermented Soy Based Product on Cardiometabolic Risk Factors
Acronym: FS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Professor of Nutrition, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 5180083
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Risk Factor; Heart Diseases; Inflammation
Keywords: Fermented Soy; Cardiovascular Disease; Inflammation; DNA Methylation
MeSH Terms: conditions — Heart Diseases; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This dietary intervention trial is a randomized, 2x2 crossover design with 24 subjects in free-living conditions.There will be a two week run-in (acclimation period), after which subjects will be randomized to receive either Q CAN powder or placebo powder for 12 weeks. Following a two week wash out period, subjects will be switched over to the alternate treatment.
Who Masked: Participant, Investigator
Masking Description: Both the participants and the investigators will not be aware of which powder is the active powder and which one is the placebo. Only the Principle Investigator will be made aware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Q CAN PLUS POWDER (Experimental): QCAN PLUS POWDER:2 pouches per day, each pouch contains(12-15gms of fermented soy powder)
  Interventions: Dietary Supplement: Q CAN PLUS
- placebo (Placebo Comparator): Sprouted brown rice protein with flavor (provided by BESO Biological Research Inc.)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Q CAN PLUS — Active powder with fermented soy , 2 pouches per day, each pouch contains 12-15 gms of fermented soy
  Arms: Q CAN PLUS POWDER
Dietary Supplement: Placebo — Sprouted brown rice protein with flavor (provided by BESO Biological Research, Inc.)
  Arms: placebo

SUMMARY:
This research study will test the effects of Q CAN PLUS powder on serum lipids, selected inflammatory and oxidative parameters and genome-wide methylation

DETAILED DESCRIPTION:
The purpose of this research study is to investigate the effects of a dietary supplement from soybeans that might help in managing heart disease. The rationale for this study is to reduce the risk factors of heart disease in high risk individuals by using soy supplements. The dietary supplement intervention trial is a randomized, 2x2 cross over design with 24 subjects in free-living conditions. There will be a two week run-in (acclimation period) after which subjects will be randomized to receive either QCAN powder or placebo powder for 12 weeks. Following a two week wash out period, subjects will be switched over(cross over) to alternate treatment. Thus, the interventions of the study will last for a total of 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 29-75 years of age
* At high risk for cardiovascular disease, i.e. with 2 or more risk factors:
* Present tobacco smoker
* Arterial hypertension (BP ≥ 140/90 mm Hg or treatment)
* LDL-cholesterol ≥ 110 mg/dl
* HDL-cholesterol ≤ 40 mg/dl
* Triglycerides ≥ 150 mg/dl
* Fasting blood glucose ≥ 110 mg/dl
* Overweight or obesity (BMI ≥ 25 kg/m2)
* Family history of premature heart disease

Exclusion Criteria:

* Uncontrolled renal, hepatic, or endocrine disease
* Abnormal blood chemistry profile
* Familial hypercholesterolemia or other genetic dyslipidemia
* Intake of lipid-lowering drugs and dietary products including plant sterols/stanols
* High Framingham risk or medical condition in which statin therapy is considered necessary by a treating physician
* Hypersensitive or allergic to soy or cellulose
* Alcohol or drug addiction or abuse
* Diabetes
* Lack of ability or interest to follow the dietary intervention

Ages: 29 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
To test the effects of Q CAN PLUS powder, on serum lipids | baseline to 7 months
  This is a composite measurement which will measure the change in the levels of serum Low Density Cholesterol, High Density Cholesterol, ApoLipoprotein A and B, APO E Allele genetic typing and triglycerides before the ingestion of QCAN PLUS powder and at 7 months after ingestion of Q CAN PLUS powder.
Inflammatory parameter | baseline to 7 months
  to test the changes in concentration of hs-CRP (highly sensitive C reactive protein) in the blood prior to ingestion of Q CAN PLUS powder and again at 7 months after ingestion of Q CAN PLUS Powder

SECONDARY OUTCOMES:
Fasting Glucose | baseline to 7 months
  to test the changes in the concentration of fasting glucose levels in the blood prior to ingestion of Q CAN PLUS powder and again after 7 months after ingestion of QCAN PLUS powder

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabate, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung SM, Haddad EH, Kaur A, Sirirat R, Kim AY, Oda K, Rajaram S, Sabate J. A Non-Probiotic Fermented Soy Product Reduces Total and LDL Cholesterol: A Randomized Controlled Crossover Trial. Nutrients. 2021 Feb 6;13(2):535. doi: 10.3390/nu13020535. PMID 33562090